CLINICAL TRIAL: NCT05581771
Title: Factors Associated With Success of Non-invasive Positive Pressure Ventilation in Patients With Amyotrophic Lateral Sclerosis: A Retrospective Cohort Study
Brief Title: Factors Associated With Success of NIPPV in ALS Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jaewon Beom, Clinical Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2210-786-107
Record Dates: First submitted 2022-10-04; First posted 2022-10-17 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: ALS
Keywords: Noninvasive positive pressure ventilation; Amyotrophic lateral sclerosis; Adherence
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective cohort study to assess the factor associated with success of non-invasive positive ventilation in ALS patients.

DETAILED DESCRIPTION:
Patients with ALS who were admitted to a tertiary hospital for initially applying non-invasive positive pressure ventilation (NIPPV). The objective of this study was to investigate factors associated with optimal NIPPV initiation and adherence, and to assess the long-term effects of NIPPV adherence in ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the El Escorial World Federation criteria for probable, or definite ALS
* Aged ≥ 19 years
* Patients who performed blood gas analysis including venous blood gas and arterial blood gas before NIPPV application.

Exclusion Criteria:

* Patients who had experience in applying the NIPPV or currently using NIPPV
* Patients who applied in outpatient settings
* Patients who did not perform blood gas analysis before NIPPV application
* Patietns who had a history of asthma or COPD,
* Patients who didn't have any record of NIPPV application time

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS patients who were admitted for applying non-invasive positive pressure ventilation initially.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Success of NIPPV | through intervention completion, with an average of 10 days
  The success of NIPPV application was defined empirically as use of ≥ 2 hours per day and the failure as use of < 2 hours for a day or conversion to invasive positive pressure ventilation via tracheostomy or refuse to apply NIPPV during hospitalization.

SECONDARY OUTCOMES:
Lenght of stay | through intervention completion, with an average of 10 days
  The length of stay (LOS) was defined as the interval between admission and hospital discharge, and calculated as the number of midnights between admission and discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Jaewon Beom, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided